CLINICAL TRIAL: NCT03147651
Title: Exercise Capacity in Patients With Cystic Fibrosis vs. Non-cystic Fibrosis Bronchiectasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 0048-15-RMB-CTIL
Record Dates: First submitted 2017-04-30; First posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Bronchiectasis
Keywords: Cystic fibrosis; exercise capacity; non-cystic fibrosis; bronchiectasis
MeSH Terms: conditions — Bronchiectasis; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cystic Fibrosis (CF) bronchiectasis: Diagnosis of Cystic Fibrosis (CF), follow up in a CF center, evidence of bronchiectasis on computed tomography (CT).
- non-Cystic Fibrosis (CF) bronchiectasis: Negative evaluation for of Cystic Fibrosis (CF), evidence of bronchiectasis on computed tomography (CT).

SUMMARY:
Introduction: Bronchiectasis is a chronic lung disease in which the underlying condition causes permanent damage to the conducting airways. Bronchiectasis is associated with considerable morbidity and poor quality of life. While cystic fibrosis (CF) is the most common cause of bronchiectasis in childhood, non-CF bronchiectasis is associated with a wide variety of disorders. CF bronchiectasis patients show reduced daily habitual physical activity and exercise capacity. Cardiopulmonary exercise test (CPET) is increasingly gaining importance in clinical medicine and considered the gold standard exercise test for assessing aerobic exercise capacity. The test objectively evaluates exercise physiological functions, may help assess morbidity and predict the outcome and mortality in different clinical circumstances and may serve as a basis for individualized exercise prescription within the limitation of the disease. Unlike CPET in CF, there is a paucity of data on exercise capacity using CPET in non- CF bronchiectasis patients, and on the implications of physical activity on non- CF bronchiectasis morbidity and mortality.

Aim: To evaluate and compare exercise capacity in CF and non-CF bronchiectasis patients.

Methods: This will be a cross-sectional retrospective/prospective study population. The retrospective study will include data analysis of patients that preformed CPET as part of their clinical evaluation. In the prospective study, patients that are scheduled to perform CPET as part of their clinical evaluation will sign (or legal guardian) informed consent prior to participation. Patients will be recruited from the exercise clinic at the Pediatric Pulmonary Institute at the Rappaport Children's Hospital. Inclusion criteria: 1. Children and adults (age >7 years, height >125cm), with CF and non CF bronchiectasis. 2. Completed a maximal CPET test according to accepted criteria; (maximal VO2 > 80% predicted, maximal heart rate > 80% predicted, acceptable RER (RER > 1.0 in children (under 18 years), RER > 1.05 for adults) or reaching a VO2 plateau..3. Evidence of bronchiectasis in computed tomography (CT).

Exclusions criteria: preforming submaximal CPET, lack of data from the exercise test, exacerbation of patient's condition within three days before the exercise evaluation, relevant related chronic diseases that affecting test results.

DETAILED DESCRIPTION:
Introduction:

Bronchiectasis is a chronic lung disease in which the underlying condition causes permanent damage to the conducting airways. Bronchiectasis is associated with considerable morbidity and poor quality of life. Patients with respiratory diseases show reduced daily functional physical ability (habitual physical activity). Reasons may be due to pulmonary limitation (in severe diseases), peripheral muscular changes or due to secondary factors such as deconditioning or overly cautious caregivers restraining patient's physical activity. Deconditioning due to reduced habitual activity leads to further reduction in exercise capacity increasing the severity of their condition. While CF is the most common cause of bronchiectasis in childhood, non-CF bronchiectasis is associated with a wide variety of disorders. The etiology for non-CF bronchiectasis include: primary ciliary dyskinesia (PCD), post infectious, aspiration, primary and secondary immunodeficiency, congenital malformation, and others. Children with CF tend to perform poorly at a moderate-intensity physical activity compared to non-CF children of same age. In the last several decades, exercise has been encouraged in CF patients to improve sputum expectoration and lung function. There is evidence that exercise in addition to respiratory physical therapy, improves lung function and reduces the rate of lung function deterioration, compared with respiratory physical therapy alone. Another study showed that an aerobic training program in children contributed to significantly higher peak aerobic capacity, activity level, and subjective quality of life than children who received a resistance training program. In conclusion, higher levels of physical activity in addition to good muscular and pulmonary functions are associated with a high aerobic capacity in cystic fibrosis.

Although the exact physiologic mechanism by which exercise improves clearing of airways secretions in CF is not entirely clear, possible explanations are attributed to increased airflow and mechanical clearing of mucus. Following physical exertion there is an increase in tidal volume and respiratory flow to meet tissue demands. Increasing peak expiratory flow (PEF) to peak inspiratory flow (PIF) ratio may help drive the mucus past the oropharynx to clear more easily. Additional benefits of exercise in patients with CF are similar to the healthy population and includes overall improvement in cardiovascular health, musculoskeletal health, and quality of life. Maximal oxygen consumption (VO2peak) serves as a strong prognosis marker associated with an approximate 8-year survival in CF patients and correlates with the number of hospital admissions due to respiratory exacerbations. There is paucity of data regarding exercise capacity in non-CF bronchiectasis.

3. Research Aim: To evaluate and compare exercise capacity in CF and non-CF bronchiectasis patients.

4. Significance: There is limited data regarding exercise capability in non-CF bronchiectasis. CPET is increasingly gaining importance in clinical medicine. The test helps the clinician objectively evaluate the physiological functions, may help predict the outcome and mortality in different clinical circumstances and may serve as a basis for creating individualized exercise prescription within the context and limitation of the disease.

5. Research Plan: Design: cross-sectional retrospective/prospective study population. The retrospective study will include data analysis of patients that preformed exercise tests as part of their clinical evaluation. In the prospective study, informed consent will be sign by the patient or legal guardian prior to participation. Setting: Outpatient clinic. The aim is to evaluate 50 patients with CF and 50 non-CF bronchiectasis patients from the exercise clinic at the Pediatric Pulmonary Institute at the Rappaport Children's Hospital.

Inclusion criteria: 1. Children and adults (age >7 years, height >125cm , with CF and non CF bronchiectasis. 2. Completed a maximal CPET test according to accepted criteria; (maximal VO2 > 80% predicted, maximal heart rate > 80% predicted, acceptable RER (RER > 1.0 in children (under 18 years), RER > 1.05 for adults) or reaching a VO2 plateau .

3. Evidence of bronchiectasis in computed tomography (CT); followed at the Pediatric Pulmonary Institute.

Exclusions criteria: preforming submaximal CPET, lack of data from the exercise test, exacerbation of patient's condition within three days before the exercise evaluation, relevant related chronic diseases that affecting test results.

The clinic has performed tests in over 1500 adolescents, children and adults, most commonly who have chronic illness such as congestive heart failure (CHD), CF, PCD, post oncological diseases, diabetes, etc.

Methods:

Age, sex, height and weight, etiology of bronchiectasis, and chest CT will be recorded. Body mass index (BMI) will be calculated. Each patient will fill a questionnaire regarding his life style and exercise capability in real life.

CPET: Following baseline measures, each patient will undergo CPET using cycle ergometer (Cosmed, Rome, Italy). Silicone face masks will be harnessed over the subject's nose and mouth to monitor the resting and exercise gas exchange measurements. Subjects are connected to electrocardiogram (ECG), saturation and blood pressure monitors. Exercise time is 8-12 minutes and total test duration is 45-60 minutes. The test is non-invasive and within the limits of the test, it is safe. The test begins with a no resistance warm up lasting 1 to 3 minutes and followed with a gradual increment in resistance adapted to the patient's functional capacities according to the examiner's free judgment and ranging 5 to 25 Watts/minute. Pulmonary function tests rest will be recorded prior to CPET and 10 minutes post exercise. The cardio-respiratory parameters measured include respiration rate (RR), heart rate by 12-lead ECG (HR), oxygen saturation (SpO2), blood pressure (BP), tidal volume (TV), minute ventilation (VE), breathing reserve (BR), oxygen consumption (VO2), VCO2 (carbon dioxide flow rejected by the ventilation system), respiratory equivalents (VE/VO2, VE/VCO2), end tidal carbon dioxide (ETCO2), anaerobic threshold (AT), oxygen pulse (O2 pulse), respiratory exchange ratio (RER) at rest, during exercise and recovery . The combination of data collected allows analysis of the subject's ability during exercise.

Spirometry: Spirometry will be performed in accordance with ATS/ERS (American Thoracic Society/ European Respiratory Society) Task Force using a KoKo spirometer (KoKo system, PDS Inc., Ferraris Cardiopulmonary System Group; Louisville, CO, USA). Each maneuver will be repeated for at least three technically acceptable; the best results were used for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of bronchiectasis on computed tomography (CT)
* Age > 7 years
* Height > 125cm
* Completed a maximal CPET test according to the accepted criteria

Exclusion Criteria:

* Preforming submaximal CPET
* Lack of data from the exercise test
* Exacerbation of patient's condition within three days before the exercise evaluation
* Related chronic diseases affecting test results

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CF and non-CF Bronchiectasis patients evaluated by CPET as part as their clinic follow up.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Oxygen Uptake (VO2) | Measured continuously during 15 minutes of the exercise test (CPET).
  Amount of oxygen consumed per amount of time.

SECONDARY OUTCOMES:
Spirometry | 5 minutes of evaluation, completed pre and post exercise test (CPET).
  Pulmonary function as assessed by spirometry.
Oxygen saturation | Measured continuously during 15 minutes of the exercise test (CPET).
  Oxygen saturation during exercise test.
Minute ventilation (VE) | Measured continuously during 15 minutes of the exercise test (CPET).
  Amount of air volume inhaled per minute of measurement.
carbon dioxide production (VCO2) | Measured continuously during 15 minutes of the exercise test (CPET).
  Amount of oxygen consumed per amount of time.

CONTACTS AND LOCATIONS:
Overall Officials: Lea Bentur, Prof., Principal Investigator — Rambam Health Care Campus
Locations (1):
- RAMBAM Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bar-Yoseph R, Ilivitzki A, Cooper DM, Gur M, Mainzer G, Hakim F, Livnat G, Schnapp Z, Shalloufeh G, Zucker-Toledano M, Subar Y, Bentur L. Exercise capacity in patients with cystic fibrosis vs. non-cystic fibrosis bronchiectasis. PLoS One. 2019 Jun 13;14(6):e0217491. doi: 10.1371/journal.pone.0217491. eCollection 2019. PMID 31194748